CLINICAL TRIAL: NCT02006121
Title: Multicentre,Parallel-group,Double-blind,Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Apomorphine sc Infusion in Parkinson's Disease Patients With Motor Complications Not Well Controlled on Medical Treatment
Brief Title: Clinical Trial of Apomorphine Subcutaneous Infusion in Patients With Advanced Parkinson's Disease
Acronym: TOLEDO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Britannia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-37527-13-0124; 2013-000980-10 (EudraCT Number)
Record Dates: First submitted 2013-11-22; First posted 2013-12-09 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; motor fluctuations; not well controlled; medical treatment; apomorphine
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apomorphine hydrochloride (Active Comparator): Apo-go® Apomorphine hydrochloride 5 mg/ml solution for infusion in pre-filled syringe
  Interventions: Drug: Apomorphine hydrochloride
- Placebo (Placebo Comparator): Placebo: saline infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine hydrochloride — Apomorphine hydrochloride 5 mg/ml solution for infusion in pre-filled syringe
  Other Names: Apo-go
  Arms: Apomorphine hydrochloride
Drug: Placebo — Sodium chloride 9 mg/ml
  Arms: Placebo

SUMMARY:
The primary objective of the trial was to investigate the efficacy of apomorphine continuous subcutaneous infusion compared to placebo in Parkinson's Disease patients with motor fluctuations not well controlled on medical treatment.

The secondary objective of the study was to investigate the safety and tolerability of apomorphine continuous subcutaneous therapy.

DETAILED DESCRIPTION:
The primary efficacy variable is the mean change in time spent "OFF" from baseline (start of blinded treatment) to the end of a 12 weeks' double-blind treatment period based on patient diaries. Patients recorded their motor symptoms in half-hour blocks as OFF, ON without dyskinesia, ON without troublesome dyskinesia, or sleeping using the Hauser Parkinson's Disease home diary.

Key secondary Endpoints (tested hierarchically):

* Change in time spent "ON without troublesome dyskinesia"
* Patient Global Impression of Change

Other Endpoints:

* Percentage of patients with response to therapy, defined as a mean OFF time reduction of at least 2 hours
* Change in oral levodopa and levodopa equivalent dose

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥30 years
* Diagnosis of idiopathic PD of >3 years' duration, defined by the UK Brain Bank criteria (with the exception of >1 affected relative being allowed), without any other known or suspected cause of Parkinsonism
* Hoehn & Yahr stage up to 3 in the ON and 2 to 5 in the OFF state
* Motor fluctuations not adequately controlled on medical treatment including levodopa which was judged by the treating physician to be optimal
* Average of OFF time > 3 hours/day based on screening and baseline diary entries with no day with < 2 hours of OFF time recorded
* Stable medication regimen, with a stable dose of levodopa administered in at least 4 intakes, for at least 28 days prior to baseline. All oral or transdermal antiparkinsonian drugs were permitted, with the exception of budipine. This regimen might include the use of levodopa/DDCI rescue medication, if this occurred up to 2 times a day, at doses of up to 200 mg levodopa/day
* Patients must be able to differentiate between the ON and OFF state and between troublesome and non-troublesome dyskinesias
* Male and female patients must be compliant with a highly effective contraceptive method (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method) during the study and for the 12-month OLP, if sexually active
* Females of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) or urine pregnancy test at screening
* Ability to accurately complete a paper diary on designated days (with assistance from caregivers, if required), recording periods when they are "ON without troublesome dyskinesia", "ON with troublesome dyskinesia", OFF, and sleeping
* Written informed consent prior to enrolment, after being provided with detailed information about the nature, risks, and scope of the clinical trial as well as the expected desirable and adverse effects of the study treatments
* Patients considered reliable and capable of adhering to the protocol, visit schedule, and medication intake according to the judgment of the investigator

Exclusion Criteria:

* History of respiratory depression
* Hypersensitivity to apomorphine or any excipients of the medicinal product
* High suspicion of other parkinsonian syndromes
* Presence of severe freezing or clinically relevant postural instability leading to falls during the ON state
* Concomitant therapy or within 28 days prior to baseline with: apomorphine pen injections; alpha-methyl dopa, metoclopramide, reserpine, neuroleptics, methylphenidate, or amphetamine; intrajejunal levodopa
* Previous use of apomorphine pump treatment
* History of deep brain stimulation or lesional surgery for PD
* Any medical condition that is likely to interfere with an adequate participation in the study, including e.g. current diagnosis of unstable epilepsy; clinically relevant cardiac dysfunction and/or myocardial infarction or stroke within the last 12 months
* Symptomatic, clinically relevant and medically uncontrolled orthostatic hypotension
* Patients with a borderline QT interval corrected for heart rate according to Bazett's formula (QTcB) of >450 msec for male and >470 msec for female at screening or history of long QT syndrome; or >450 msec absolute duration
* Clinically relevant hepatic dysfunction (total bilirubin >2.0 mg/dL, alanine transaminase [ALT] and aspartate transaminase [AST] >2 times the upper limit of normal)
* Clinically relevant renal dysfunction (serum creatinine >2.0 mg/dL)
* Pregnant and breastfeeding women
* Clinically relevant cognitive decline, defined as MMSE ≤24 or according to Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria for dementia
* Active psychosis or history of at least moderate psychosis in the past year, or with medically uncontrolled severe depression; very mild illusions or hallucinations in the sense of "feelings of passage or presence" with fully retained insight are not an exclusion criterion
* Known history of melanoma
* Any investigational therapy in the 4 weeks prior to randomization
* History or current drug or alcohol abuse or dependencies

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina Katzenschlager, Doz. Dr., Principal Investigator — Donauspital KH SMZ Ost, Neurologie
Locations (20):
- Austria (3):
  - Medizinische Universität Graz / Univ. Klinik für Neurologie, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Donauspital / SMZ-Ost, Abteilung für Neurologie, Sekretariat (Stock 1, Ebene 4), Vienna
- Bispebjerg University Hospital, Movement Disorder Centre, Copenhagen, Denmark
- France (3):
  - CHRU Clermont- Ferrand Gabriel-Montpied, Clermont-Ferrand
  - CHU de Rennes, Hôpital Pontchaillou, Rennes
  - CHU Toulouse, Hôpital Purpan, Centre d'Investigation Clinique, Toulouse
- Germany (4):
  - Neurologisches Fachkrankenhausfür Bewegungsstörungen / Parkinson, Beelitz-Heilstätten
  - Klinikum Bremerhaven-Reinkenheide gGmbH, Neurologische Klinik, Bremerhaven
  - Paracelsus Elena-Klinik Kassel, Kassel
  - Schön Klinik München Schwabing / Neurologie und Klinische Neurophysiologie, München
- Netherlands (3):
  - Universitair Medisch Centrum, Groningen
  - Atrium MC parkstad, Heerlen
  - Erasmus MC, Rotterdam
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
- United Kingdom (4):
  - The Walton Centre Nhs Foundation Trust, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - St George's Heathcare NHS Trust, London
  - Newcastle University, Clinical Ageing Research Unit (CARU), Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katzenschlager R, Poewe W, Rascol O, Trenkwalder C, Deuschl G, Chaudhuri KR, Henriksen T, van Laar T, Lockhart D, Staines H, Lees A. Long-term safety and efficacy of apomorphine infusion in Parkinson's disease patients with persistent motor fluctuations: Results of the open-label phase of the TOLEDO study. Parkinsonism Relat Disord. 2021 Feb;83:79-85. doi: 10.1016/j.parkreldis.2020.12.024. Epub 2021 Jan 12. PMID 33486139
- [Derived] Katzenschlager R, Poewe W, Rascol O, Trenkwalder C, Deuschl G, Chaudhuri KR, Henriksen T, van Laar T, Spivey K, Vel S, Staines H, Lees A. Apomorphine subcutaneous infusion in patients with Parkinson's disease with persistent motor fluctuations (TOLEDO): a multicentre, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2018 Sep;17(9):749-759. doi: 10.1016/S1474-4422(18)30239-4. Epub 2018 Jul 25. PMID 30055903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Blinded treatment was administered over 12 weeks after which patients could choose to enrol in a 12-month open-label phase. Early switching to the open-label phase was permitted for lack of efficacy in the double-blind phase.
Groups:
- Apomorphine Hydrochloride: Apo-go® Apomorphine hydrochloride 5 mg/ml solution in 10 mL pre-filled syringes for continuous infusion during the waking day using a Cane CRONO APO-Go® infusion pump. Hourly flow rate adjusted in increments of 0.5-1.0 mg/hour/day during titration to reach the patient's individualized required dose in a range of 3-8 mg/hour for 14-18 hours per day.
  Concomitant medications were reduced/discontinued in the following order: dopamine agonists, MAO-B inhibitors, COMT inhibitors, levodopa dose then frequency.
- Placebo: Blinded Placebo: saline infusion; Open Label, placebo switched to apomorphine infusion.
  Blinded phase: Sodium chloride 9 mg/ml continuous infusion during the waking day using a Cane CRONO APO-Go® infusion pump. Hourly flow rate adjusted in increments of 0.5-1.0 mg/hour/day during titration to reach the patient's individualized required dose in a range of 3-8 mg/hour for 14-18 hours per day.
  Concomitant medications were reduced/discontinued in the following order: dopamine agonists, MAO-B inhibitors, COMT inhibitors, levodopa dose then frequency.
  Open Label phase: as per apomorphine arm
Period: Double Blind Phase
Arm/Group | Apomorphine Hydrochloride | Placebo
Started | 54 | 53
Completed | 42 (Early switching to open label: 1 for lack of efficacy, 1 could not tolerate 3 mg/hour minimum rate) | 29 (16 placebo-treated patients early switched to open label phase due to lack of efficacy)
Not Completed | 12 | 24
Not completed — Adverse Event | 6 | 0
Not completed — Lack of Efficacy | 1 | 16
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Non-compliance with study drug | 1 | 3
Not completed — Minimum infusion rate poorly tolerated | 1 | 0
Not completed — Inconvenience of infusion system | 0 | 1
Period: Open Label Phase
Arm/Group | Apomorphine Hydrochloride | Placebo
Started | 84 (From Apo: 38 completers and 2 early switched; From Placebo: 28 completers and 16 early switched) | 0 (No patients received placebo in the open label phase)
Completed | 59 (30 who continued on apomorphine from blinded phase, 29 who switched to apomorphine from placebo) | 0
Not Completed | 25 | 0
Not completed — Adverse Event | 15 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Non-compliance with study drug | 3 | 0

BASELINE CHARACTERISTICS:
Population: Demographic Characteristics displayed for mITT population
Groups:
- Placebo: Placebo: saline infusion Sodium chloride 9 mg/ml
- Total: Total of all reporting groups
Arm/Group | Apomorphine Hydrochloride | Placebo | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.58 (9.32) | 63.00 (8.32) | 63.29 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Daily OFF Time From Baseline (Start of Blinded Treatment) to the End of Double-blind Phase (Visit 10) Based on Patient Diaries Using MMRM mITT Population
Description: The least squares mean reduction (improvement) in OFF time as reported by the patient using the Hauser Parkinson's disease home diary. Patients categorised their motor symptoms into OFF, ON with dyskinesia, ON without troublesome dyskinesia or sleeping using half hour blocks over 24 hours. Daily OFF time was computed from the average of valid motor diaries from the two days preceding each visit. Correct diary completion was evaluated during screening and observed by the investigator to ensure patients could categorise their motor symptoms correctly. A diary was considered valid if no more than 4 half-hour periods were either absent or duplicated. There were no invalid diaries at Baseline or Week 12.
Time Frame: Baseline and 12 weeks
Population: All randomised patients excluding those who had major protocol deviations who received at least one dose of trial medication during the course of the trial and for whom any post-baseline efficacy assessment is available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Apomorphine Hydrochloride | Placebo
Number analyzed (Participants) | 53 | 52
Hours | -2.61 [-3.43 to -1.80] | -0.75 [-1.66 to 0.16]
Statistical Analysis 1: Comparison: Apomorphine Hydrochloride vs Placebo; Test type: Superiority; p = 0.0047, Mixed Models Analysis

2. Secondary Outcome: Mean Change in Daily Time Spent "ON Without Troublesome Dyskinesia" From Baseline to the End of the Double-blind Phase (Visit 10), Based on Patient Diaries Using MMRM mITT Population
Description: The least squares mean change in "ON time without troublesome dyskinesia" as reported by the patient using the Hauser Parkinson's disease home diary. Each half hour of the day categorised as OFF, ON with dyskinesia, ON without troublesome dyskinesia or asleep. "ON time without troublesome dyskinesia" measures good ON time for a Parkinson's disease patient.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Apomorphine Hydrochloride | Placebo
Number analyzed (Participants) | 53 | 52
Hours | 2.90 [2.07 to 3.73] | 0.85 [-0.09 to 1.78]
Statistical Analysis 1: Comparison: Apomorphine Hydrochloride vs Placebo; Test type: Superiority; p = 0.0022, Mixed Models Analysis

3. Secondary Outcome: Patient Global Impression of Change (PGIC), Using the mITT Population
Description: PGIC is a self-administered questionnaire measuring personal general state of health on a 7-point rating scale. The 7 ordinal categories from which patients must choose are 'very much improved', 'much improved', 'minimally improved', 'no change', 'minimally worse', 'much worse', and 'very much worse. Results are presented as the % of patients who reported at least minimal improvement in general health status at week 12 compared to Baseline. A Wilcoxon range sum test was performed to test for treatment differences from baseline to end of 12 weeks' treatment period.
Time Frame: Baseline and 12 weeks
Population: All randomised patients excluding those who had major protocol deviations who received at least one dose of trial medication during the course of the trial and for whom any post-baseline efficacy assessment is available and who completed the PGIC questionnaire
Measure: Number; unit: % of participants
Arm/Group | Apomorphine Hydrochloride | Placebo
Number analyzed (Participants) | 43 | 34
% of participants | 79.1 | 23.5
Statistical Analysis 1: Comparison: Apomorphine Hydrochloride vs Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mean Change in Oral Levodopa Dose From Baseline to Visit 10 Using MMRM for the mITT Population
Description: The least squares mean change in oral levodopa dose from Baseline to Visit 10 (week 12) was calculated excluding 3 centres who declined to participate in collecting the necessary details of PRN use of levodopa.
Time Frame: Baseline and 12 weeks
Population: All patients who received at least one dose of randomized study medication and had at least one post-baseline observation for the primary endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Apomorphine Hydrochloride | Placebo
Number analyzed (Participants) | 41 | 32
mg | -242.09 [-346.58 to -137.61] | -76.46 [-185.17 to 32.25]
Statistical Analysis 1: Comparison: Apomorphine Hydrochloride vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis

5. Secondary Outcome: Mean Change in Levodopa Equivalent Dose From Baseline to Visit 10 (Week 12) Using MMRM in the mITT Population
Description: Levodopa equivalent dose is an indication of the burden of medication taken to control symptoms of Parkinson's disease with all medications other than levodopa itself being converted to a calculated levodopa dose using the methodology published by Tomlinson et al, 2010. The computation of LED excludes the study drug.
Time Frame: Baseline and 12 weeks
Population: All randomized patients treated at least once with study medication and who had at least one post-baseline observation for the primary endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Apomorphine Hydrochloride | Placebo
Number analyzed (Participants) | 49 | 48
mg | -502.02 [-626.45 to -377.60] | -150.87 [-280.14 to -21.59]
Statistical Analysis 1: Comparison: Apomorphine Hydrochloride vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the double-blind and open label phases of the study. 98 patients were exposed to at least one dose of apomorphine with a cumulative person time of 4081 weeks of exposure. The range of exposure to apomorphine was 37-464 days (mean 397 days). In addition, 53 patients (44 of whom went onto apomorphine in the open label phase) were exposed to placebo treatment in the double blind phase with a maximum 12 weeks of exposure.
Arm/Group | Apomorphine Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/53
Serious Adverse Events (participants affected / at risk) | 23/98 | 2/53
Other Adverse Events (participants affected / at risk) | 94/98 | 30/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apomorphine Hydrochloride (N=98) | Placebo (N=53)
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Infusion site cellulitis (Infections and infestations) | 2 | 0
Eosinophil count decreased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Blood disorder (Blood and lymphatic system disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
On Off phenomenon (Nervous system disorders) | 1 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Device difficult to use (Product Issues) | 1 | 0 — Patient's carer admitted to hospital, he could not use pump and was admitted in OFF state. Retrained on pump and discharged on treatment
Paranoia (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep brain stimulation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apomorphine Hydrochloride (N=98) | Placebo (N=53)
Infusion site nodule (General disorders) | 46 | 0
Infusion site erythema (General disorders) | 15 | 2
Infusion site haematoma (General disorders) | 8 | 5
Fatigue (General disorders) | 6 | 1
Oedema peripheral (General disorders) | 7 | 0
Infusion site pruritus (General disorders) | 5 | 0
Somnolence (Nervous system disorders) | 19 | 2
Headache (Nervous system disorders) | 10 | 2
Dyskinesia (Nervous system disorders) | 14 | 0
Dizziness (Nervous system disorders) | 11 | 2
Nausea (Gastrointestinal disorders) | 20 | 5
Vomiting (Gastrointestinal disorders) | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 1
Insomnia (Psychiatric disorders) | 13 | 1
Hallucination, visual (Psychiatric disorders) | 6 | 2
Sleep disorder (Psychiatric disorders) | 6 | 1
Hallucination (Psychiatric disorders) | 5 | 0
Nasopharyngitis (Infections and infestations) | 7 | 3
Urinary tract infection (Infections and infestations) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Orthostatic hypotension (Vascular disorders) | 6 | 1
Eosinophilia (Blood and lymphatic system disorders) | 5 | 0
Electrocardiogram QT prolonged (Investigations) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No